CLINICAL TRIAL: NCT05385757
Title: Uveitis in Childhood Prospective National Cohort Study
Brief Title: UNICORNS: Uveitis in Childhood Prospective National Cohort Study
Acronym: UNICORNS
Status: Active, not recruiting | Type: Observational
Sponsor: Institute of Child Health (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 258638
Record Dates: First submitted 2020-10-16; First posted 2022-05-23 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Uveitis
Keywords: Quality of life; Child; Prospective Cohort; Vision
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Saliva, Stool, Tears and Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Childhood Uveitis: Children <18 years old newly diagnosed with non-infectious uveitis

SUMMARY:
Childhood uveitis (inflammation inside the eye) is an uncommon disorder that carries the risk of blindness. Inadequate treatment of active inflammation has been shown to be related to a poor outcome. There has been no population-based, prospective longitudinal study of all-cause childhood uveitis, with resultant limitations in the evidence base used to counsel affected families, balance treatment decisions, or plan further research. The aim of the study is to describe the characteristics of childhood-onset uveitis and describe outcomes. The investigators shall also aim to identify the socio-demographic, clinical, biological and treatment-related determinants of outcome. Early (1-2 years following diagnosis) outcomes will be described in the first instance: However, through the creation of a national inception cohort, the investigators shall enable longer-term studies of outcome for affected children and families. There will be no change to routine clinical care.

DETAILED DESCRIPTION:
Background:

Childhood uveitis descriptive term for a group of rare inflammatory eye disease, which are typically chronic, relapsing-remitting in nature, and of uncertain aetiology (idiopathic). Visual loss occurs due to structural damage caused by uncontrolled inflammation. Understanding of the determinants of long-term outcome is limited, particularly the predictors of therapeutic response or how to define disease control.

Aims:

To describe disease natural history and outcomes amongst a nationally representative group of children with non-infectious uveitis, describe the impact of disease course on quality of life for both child and family, and identify determinants of adverse visual, structural and developmental outcomes.

Methods:

UNICORNS is a prospective longitudinal multicentre cohort study of children newly diagnosed with uveitis about whom a core minimum clinical dataset will be collected. Participants and their families will also complete patient-reported outcome measures (PROMS) at study entry and annually from recruitment.

PROMS collected at baseline are:

* Strength and Difficulties Questionnaire (SDQ): this is to screen the emotional and behavioural aspects of the participants' lives
* Child Health Utility 9D (CHU9D): generic preference based measure of health related quality of life
* Children's Sleep Habits Questionnaire (CHSQ): this evaluates incidence of behaviours linked with typical paediatric sleep difficulties
* 100-mm General Evaluation (GE): visual analogue score 100mm long used to capture overall perception of the burden of disease

PROMS collected at year 1 and annually (subject to investigations of instrument redundancy) are:

* Child Health Utility 9D (CHU9D): generic preference based measure of health related quality of life
* 100-mm General Evaluation (GE): visual analogue score 100mm long used to capture overall perception of the burden of disease
* Paediatric Quality of life Score (PedsQL): a brief questionnaire used to evaluate health related quality of life in children
* Vision related quality of life metric - Children and Young People (VQoL_CYP): these instruments captures the functional and broader impacts of living with a visual disability The association of patient (child- and treatment- dependent) characteristics with outcome will be investigated using logistic and ordinal regression models which incorporate adjustment for within-child correspondence between eyes for those with bilateral disease and repeated outcomes measurement.

Discussion:

Through this population based, prospective longitudinal study of childhood uveitis, the investigators will describe the characteristics of childhood onset disease. Early (1-2 years following diagnosis) outcomes will be described in the first instance, and through the creation of a national inception cohort, longer term studies of outcome for affected children and families will be enabled.

ELIGIBILITY:
Inclusion Criteria:

* Children newly diagnosed with uveitis (within previous 6 months)
* Age < 18years

Exclusion Criteria:

* Uveitis due to malignancy
* Uveitis due to ocular trauma (including iatrogenic, ie intraocular surgery)
* Uveitis due to confirmed ocular infection
* Children with developmental disorders or impairments which prevent their self-report of their function level or quality of life

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children those aged under 18 years old (at diagnosis) who are newly diagnosed with uveitis newly diagnosed with uveitis (within previous 6 months)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular complications | Up to 3 years
  New incident of sight threatening ocular complications, including glaucoma, cataract and macular oedema
Pediatric Quality of Life Inventory Score | Up to 3 years
  Quality of life (patient reported outcomes) using Pediatric Quality of Life Inventory (PedsQL) in which items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL (Health-Related Quality of Life)

SECONDARY OUTCOMES:
Corticosteroid exposure | Up to 3 years
  Total prescribed topical and systemic corticosteroid burden
Attainment of disease control | Up to 3 years
  Number of children achieving absolute control defined as absence of inflammation Relative control defined as the absence of inflammation greater than 0.5 The lowest grade of inflammation, with the use of less than one drop of topical corticosteroid
Health Utility | Up to 3 years
  Child Health Utility Metric (CHU9D), with scores ranging from 0.33 (worst health state) to 1.00 (best health state)
Change in Pediatric Quality of Life Inventory Score | Over one year from baseline to year one
  Change in child reported quality of life using Pediatric Quality of Life Inventory (PedsQL) in which items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL (Health-Related Quality of Life), and a change of greater than 5 is clinically meaningful

CONTACTS AND LOCATIONS:
Overall Officials: Ameenat L Solebo, Principal Investigator — University College London (UCL) Great Ormond Street Institute of Child Health
Locations (31):
- United Kingdom (31):
  - Belfast Royal Victoria Hospital NHS Foundation Trust, Belfast
  - Birmingham Women's and Children's Hospital NHS Foundation Trust, Birmingham
  - Royal Bournemouth Christchurch Hospitals NHS Foundation Trust, Bournemouth
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Cambridge University Hospital NHS Foundation Trust, Cambridge
  - Cardiff and Vale University Health Board Hospitals, Cardiff
  - Mid Essex Hospital Trust, Chelmsford
  - Ninewells Hospital, Dundee
  - Princess Alexandra Eye Pavilion, Edinburgh
  - Royal Children's Hospital, Glasgow
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth
  - Hull University Teaching Hospitals NHS Trust, Hull
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Alder Hey Hospital NHS Foundation Trust, Liverpool
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Royal Free London NHS Foundation Trust, London
  - St Thomas' Hospital, London
  - Great Ormond Street Hospital NHS Foundation Trust, London
  - Maidstone and Tunbridge Wells NHS Trust, Maidstone
  - Manchester University NHS Foundation Trust, Manchester
  - Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Sussex Eye Hospital and Royal Alexandra Children's Hospital, Redhill
  - Sheffield Children's Hospitals NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea
  - Royal London Hospital, Whitechapel
  - York Teaching Hospital NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: No
Authorised collaborators will be granted access to aggregated anonymised data, following review of their research protocol study PI and Co-Is. Data and material transfer agreements will be required to be completed, in order to ensure regulatory compliance and that the interests of the participants are upheld and respected throughout.

REFERENCES:
- [Background] Kellett S, Rahi JS, Dick AD, Knowles R, Tadic V, Solebo AL. UNICORNS: Uveitis in childhood prospective national cohort study protocol. F1000Res. 2023 Aug 30;9:1196. doi: 10.12688/f1000research.26689.2. eCollection 2020. PMID 38435080
- See also: Study Website — http://www.ucl.ac.uk/child-health/unicorns
- See also: Study Video — http://www.youtube.com/channel/UCRkMbO7q5sN8M_0RtggBDyQ

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT05385757/Prot_SAP_000.pdf